CLINICAL TRIAL: NCT05932446
Title: A Single Dose Study to Assess the Pharmacokinetics of 2 Formulations of LY3819469 in Healthy Participants
Brief Title: A Study to Compare Two Formulations of LY3819469 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 18730; J3L-MC-EZEE (Other: Eli Lilly and Company)
Record Dates: First submitted 2023-06-28; First posted 2023-07-06 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LY3819469 (Reference) (Experimental): LY3819469 administered subcutaneously (SC).
  Interventions: Drug: LY3819469
- LY3819469 (Test) (Experimental): LY3819469 administered SC.
  Interventions: Drug: LY3819469

INTERVENTIONS:
Drug: LY3819469 — Administered SC.

SUMMARY:
The main purpose of this study is to assess two formulations of LY3819469 based on the amount that gets into the blood stream and how long it takes the body to get rid of it, when given to healthy participants. The information about any adverse effects experienced will be collected and the tolerability of LY3819469 will also be evaluated.

Screening is required within 28 days prior to the enrolment. For each participant, the total duration of the clinical trial will be about 17 weeks including screening and follow-up periods.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants who are overtly healthy as determined by medical evaluation
* Have a body mass index (BMI) in the range of 18.5 to 35.0 kilogram per square meter (kg/m²), inclusive at the time of screening
* Are male or women not of childbearing potential

Exclusion Criteria:

* Have a history or presence of an underlying disease, or surgical, physical, medical, or psychiatric condition that could affect interpretation of study data
* Have any abnormality in the 12-lead electrocardiogram (ECG)
* Are heavy alcohol drinkers or heavy cigarette smokers
* Have participated, within the last 30 days, in a clinical study involving an investigational product. If the previous investigational product has a long half-life, 5 half-lives, or 30 days, whichever is longer, should have passed prior to CRU admission
* Have lost or donated blood of more than 450 mililitres (mL) within 3 months

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2023-06-30 (Actual); Primary Completion 2023-11-07 (Actual); Study Completion 2023-11-07 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve From Time Zero to the Last Timepoint with Measurable Concentration (AUC[0-tlast]) of LY3819469 | Predose on day 1 up to postdose on day 85
  PK: AUC[0-tlast] of LY3819469
PK: Area Under the Concentration Versus Time Curve From Time Zero to Infinity (AUC[0-∞]) of LY3819469 | Predose on day 1 up to postdose on day 85
  PK: AUC[0-∞] of LY3819469
PK: Maximum Observed Concentration (Cmax) of LY3819469 | Predose on day 1 up to postdose on day 85
  PK: Cmax of LY3819469

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Lilly Centre for Clinical Pharmacology, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dimitriadis K, Theofilis P, Iliakis P, Pyrpyris N, Dri E, Sakalidis A, Soulaidopoulos S, Tsioufis P, Fragkoulis C, Chrysohoou C, Tsiachris D, Tsioufis K. Management of dyslipidemia in coronary artery disease: the present and the future. Coron Artery Dis. 2024 Sep 1;35(6):516-524. doi: 10.1097/MCA.0000000000001375. Epub 2024 Apr 29. PMID 38682459